CLINICAL TRIAL: NCT07262697
Title: Comparison of High-intensity Laser Therapy and Low-Level Laser Therapy in Patients With Non-specific Neck Pain
Brief Title: Laser Therapy for Patients With Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Mohammad Moustafa Aldosoukki Hegazy, Assisstant professor, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHPT/022/041
Record Dates: First submitted 2025-11-18; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain; Non Specific Neck Pain
Keywords: laser; neck pain; neck disability
MeSH Terms: conditions — Neck Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: th
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HILT (Experimental): The first phase consisted of rapid manual scanning, delivering a total energy of 1000 J/cm². During the second phase, HILT was applied to eight trigger points, with four applications per point, continuing until pain reduction reached approximately 70-80%; a total of 200 J was delivered in this phase. The final phase was performed with slow manual scanning with the same parameters as the initial phase. The complete HILT procedure lasted around 30 minutes, with a total energy dose of approximately 2050 J (19).
  Interventions: Other: HILT; Other: CONTROL
- LLLT (Experimental): LLLT sessions were carried out using the diode laser device (Chattanooga Group, USA) of gallium-aluminum-arsenide (GaAlAs, infrared laser) with an 850 nm wavelength, 800 mW power, and constant wave with 1 cm spot size was utilized for the treatment procedures. The laser probe was positioned directly on specific points along the cervical spine while the participant's head remained in a neutral position. Each point was treated for 2 minutes. A total of eight points were marked bilaterally over the trapezius and sternocleidomastoid muscles, covering an area of 24 cm². The total treatment duration was 18 minutes, with an energy dose of 2 J/cm² applied to each point (20).
  Interventions: Other: LLLT; Other: CONTROL
- CONTROL (Active Comparator): The home program involved stretching exercises for levator scapulae and upper trapezius, strengthening exercises for neck extensors, and scapular stabilizer exercises. Each exercise was executed with a 5-second hold and 10 repetitions per set, for a total of three sets repeated three times per week for 10 weeks.
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: HILT — The first phase consisted of rapid manual scanning, delivering a total energy of 1000 J/cm². During the second phase, HILT was applied to eight trigger points, with four applications per point, continuing until pain reduction reached approximately 70-80%; a total of 200 J was delivered in this phase. The final phase was performed with slow manual scanning with the same parameters as the initial phase. The complete HILT procedure lasted around 30 minutes, with a total energy dose of approximately 2050 J (19).
  Other Names: Home program
  Arms: HILT
Other: LLLT — The laser probe was positioned directly on specific points along the cervical spine while the participant's head remained in a neutral position. Each point was treated for 2 minutes. A total of eight points were marked bilaterally over the trapezius and sternocleidomastoid muscles, covering an area of 24 cm². The total treatment duration was 18 minutes, with an energy dose of 2 J/cm² applied to each point (20).
  Other Names: HOME PROGRAM
  Arms: LLLT
Other: CONTROL — The home program involved stretching exercises for levator scapulae and upper trapezius, strengthening exercises for neck extensors, and scapular stabilizer exercises. Each exercise was executed with a 5-second hold and 10 repetitions per set, for a total of three sets repeated three times per week for 10 weeks.

SUMMARY:
Background and Purpose: Neck pain is widespread and stands as the sixth most common cause of disability globally. While laser therapy has been used for many years to treat non-specific neck pain (NNP), there is still a shortage of research directly comparing different laser modalities. The aim of this study was to evaluate and compare the therapeutic effectiveness of low-level laser therapy (LLLT) and high intensity laser therapy (HILT) in managing NNP.

Methods: sixty patients diagnosed with NNP were equally randomized into three groups. HILT group received 10 weeks of HILT, LLLT group received 10 weeks of LLLT and a control group that received a home program. Outcome measures were evaluated at baseline and after the intervention period and included pain intensity, neck disability, active cervical range of motion (ROM), and quality of life.

DETAILED DESCRIPTION:
Study Design This study was designed as randomized comparative trial. The study procedures were conducted in the electrotherapy laboratory in the Department of Rehabilitation and Health Sciences, Prince Sattam Bin Abdulaziz University, Al-Kharj, Saudi Arabia between March 2023 and April 2024. The study involved recruitment of 75 subjects from the university hospital and local clinics. Initial evaluation was performed by an orthopedist. The study sample included participants diagnosed with chronic non-specific neck pain (NNP) according to clinical and radiological tests. Study subjects were randomly assigned to one of three groups high intensity laser therapy (HILT) group, low-level laser therapy (LLLT) group, and a control group. The HILT group subjects underwent 10 weeks of HILT in addition to a home exercise program while the LLLT group subjects underwent 10 weeks of LLLT in addition to a home exercise program. The third group was a control group where group subjects performed only a home exercise program and did not receive laser therapy. The use of analgesics or nonsteroidal anti-inflammatory medications was not allowed during the intervention period (17).

The randomization process was conducted using SPSS statistical software, following a 1:1 allocation ratio and stratified by center, with random block sizes of four to ensure balanced distribution. An independent researcher, who was not involved in recruiting participants or delivering the interventions, generated the randomization sequence. Group assignments were recorded on numbered cards and sealed in opaque envelopes by this independent researcher. These envelopes were later opened by the intervention researchers, who administered the respective treatment according to group allocation.

Blinding was maintained throughout the study. All participants were unaware of their assigned group, ensuring subject blinding. Although the therapists delivering the treatments knew which group participants belonged to, they were blinded to the specific laser parameters, as these settings were predetermined by an independent researcher. The therapists' role was limited to implementing standardized treatment protocols without access to detailed device settings. Furthermore, all outcome evaluations were performed by an assessor who was blinded to group allocation, thereby minimizing assessment bias and maintaining the integrity of the study's double-blind design.

ELIGIBILITY:
Inclusion Criteria:

* chonic neck pain lasting more than 30 days with no evidence of foraminal compression;
* age 18 years or older;
* experiencing considerable pain, stiffness, or discomfort localized to the neck area, without associated numbness or radiation of pain to the upper limbs;
* a visual analog scale (VAS) pain rating of 3 or above;
* no therapeutic intervention within the last month

Exclusion Criteria:

* Previous cervical spine trauma or surgery;
* significant cervical disc prolapse, cervical nerve root compression or spinal cord manifestations;
* history of severe and frequent migraines, fibromyalgia, shoulder diseases, rheumatic or rheumatoid diseases, severe osteoporosis, mental illnesses, significant spinal deformities, or serious cardiovascular, pulmonary, or neurological diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 10 weeks
  VAS is a reliable tool for measuring pain intensity. Each participant was asked to mark a point on a 10 cm line corresponding to the severity of their pain, with scores ranging from 0 to 10-where 0 indicates no pain and 10 represents the most severe pain. Previous research has demonstrated that the VAS is a reliable and valid tool for assessing the intensity of neck pain

SECONDARY OUTCOMES:
Active ROM of the cervical spine | 10 weeks
  A universal goniometer was employed to quantify the angle of motion in each direction. Each movement was measured three times to ensure consistency, and the mean of the three readings was recorded as the final value. This standardized method minimizes measurement error and improves reproducibility. Previous studies have reported that cervical active ROM assessment using a goniometer provides excellent intra- and inter-rater reliability, making it a valid and dependable tool for evaluating neck mobility (23).
Functional disability | 10 weeks
  The Neck Disability Index (NDI) was employed to assess functional disability in the study participants. This instrument consists of 10 items divided into two domains: neck pain-related symptoms and the capacity to carry out daily activities. Each item is scored from 0 to 5, yielding a maximum total score of 50, with higher scores indicating greater cervical functional impairment (24). The NDI was expressed as a percentage of disability, determined by the formula (total score/50 × 100). The NDI has good internal consistency and test-retest reliability
SF-36 Quality of life | 10 weeks
  The SF-36 consists of 36 items that assess both physical and mental health, allowing participants to rate their perceived health status on a scale from 0 to 100, where 0 indicates the poorest health and 100 indicates the best possible health (26). This questionnaire provides a reliable measure of two distinct domains: physical and mental health (27).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Hegazy, Al Kharj, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ezzati K, Laakso EL, Saberi A, Yousefzadeh Chabok S, Nasiri E, Bakhshayesh Eghbali B. A comparative study of the dose-dependent effects of low level and high intensity photobiomodulation (laser) therapy on pain and electrophysiological parameters in patients with carpal tunnel syndrome. Eur J Phys Rehabil Med. 2020 Dec;56(6):733-740. doi: 10.23736/S1973-9087.19.05835-0. Epub 2019 Nov 18. PMID 31742366
- [Background] Alayat MSM, Alshehri MA, Shousha TM, Abdelgalil AA, Alhasan H, Khayyat OK, Al-Attar WS. The effectiveness of high intensity laser therapy in the management of spinal disorders: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2019;32(6):869-884. doi: 10.3233/BMR-181341. PMID 30932879